CLINICAL TRIAL: NCT02320097
Title: A Study of the Impact of Head Position on Foot Pressure in Stance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5899
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Study the Impact of Head Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foot pressure measurement (Other): The subject stands on the platform, with the heels and buttocks touching a vertical plane and the head held freely. The subject then moves his/her head backwards so that it touches the vertical plane. Next, he/she turns the head to the right and then towards the left. Each of these positions is maintained for 2 minutes.
  The platform's sensors measure the anteroposterior foot pressure distribution during the various acquisitions.
  Interventions: Other: Foot pressure measurement

INTERVENTIONS:
Other: Foot pressure measurement — Description of the foot pressure measurement:
  The subject stands on the platform, with the heels and buttocks touching a vertical plane and the head held freely. The subject then moves his/her head backwards so that it touches the vertical plane. Next, he/she turns the head to the right and then towards the left. Each of these positions is maintained for 2 minutes.
  The platform's sensors measure the anteroposterior foot pressure distribution during the various acquisitions.

SUMMARY:
When examining a subject in quiet stance from the side, the leg segment is usually seen to be oriented upwards and forwards by about 5°; the knee may be flexed by a few degrees, the shoulders are behind the great trochanter and the head is held forwards. The forward head position moves the center of gravity forwards and thus may increase pressure under the forefoot. Conversely, moving the head backwards should be accompanied by an increase in pressure under the heel and thus decreased pressure under the forefoot.

The study's objective is to study the influence of alignment of the head with the back (i.e. a rearward head position) and head rotation on the foot pressure distribution (measured using a foot pressure platform).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30
* Social security coverage
* Ability to understand the study's objectives, procedures and risks and to provide informed, written consent

Exclusion Criteria:

* Past or concomitant infectious or cancerous diseases of the spine
* Vertebral osteosynthesis
* Acute neck or arm pain
* Limb trauma in the previous 12 months
* Acute leg pain
* Neuropathic disease or the sequelae of neuropathic disease of the legs
* Myasthenia gravis
* Central nervous system disorders
* Inner ear problems
* Subjects under legal guardianship
* Known pregnancy
* Simultaneous participation in another biomedical research study of a drug or medical device.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The foot pressure in g/cm2 and the anteroposterior pressure distribution, measured using a foot pressure platform. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mutter Catherine, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg

REFERENCES:
- [Result] Nisand M, Callens C, Destieux C, Dyer JO, Chanson JB, Sauleau E, Mutter C. Baropodometric quantification and implications of muscle coactivation in the lower limbs caused by head movement: A prospective study. J Bodyw Mov Ther. 2020 Jan;24(1):228-234. doi: 10.1016/j.jbmt.2019.05.014. Epub 2019 May 15. PMID 31987549